CLINICAL TRIAL: NCT03388515
Title: A Randomized, Double-blinded, Placebo-controlled, Single-dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SSS11 Administered Intravenously in Healthy Volunteers.
Brief Title: A Study to Assess the Safety and Tolerability of SSS11 in Healthy Subjects.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSS11
Record Dates: First submitted 2017-12-05; First posted 2018-01-03 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2017-09

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SSS11, 1.5mg (Experimental): SSS11, 1.5mg, iv, single dose at Day 1;
  Interventions: Biological: SSS11; Other: placebo
- SSS11, 3.0mg (Experimental): SSS11, 3.0mg, iv, single dose at Day 1;
  Interventions: Biological: SSS11; Other: placebo
- SSS11, 6.0mg (Experimental): SSS11, 6.0mg, iv, single dose at Day 1;
  Interventions: Biological: SSS11; Other: placebo
- SSS11, 12.0mg (Experimental): SSS11, 12.0mg, iv, single dose at Day 1;
  Interventions: Biological: SSS11; Other: placebo
- SSS11, 24.0mg (Experimental): SSS11, 24.0mg, iv, single dose at Day 1;
  Interventions: Biological: SSS11; Other: placebo

INTERVENTIONS:
Biological: SSS11 — IV infusion for 60 min.
  Other Names: pegsiticase
Other: placebo — IV infusion for 60 min.

SUMMARY:
SSS11 is pegsiticase consisting of a recombinant uricase conjugated to multiple 20kDa PEG molecules. The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of single dose SSS11 administered intravenously in healthy volunteers.

DETAILED DESCRIPTION:
Objectives:

Primary:

• To assess the safety, tolerability of single dose SSS11 in healthy subjects

Secondary:

• To assess the pharmacokinetics, pharmacodynamics and immunogenicity of SSS-11 in healthy subjects

Enrollment and Number of Arms (planned):

40 subjects will be assigned into 5 dosing cohorts (1.5, 3, 6, 12 and 24mg) with 5-10 subjects each.

Original primary outcome Measures:

Safety: Physical exam，ECG，Clinical laboratory tests，AE，SAE Tolerance assessment：MDT，DLT

Original secondary outcome Measures:

pharmacokinetics: Cmax, Tmax, AUC, CL, Vd, t1/2 pharmacodynamics: level of serum uric acid Immunogenicity ：anti-SSS11, anti-uricase and anti-PEG antibodies

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-45 years of age at time of consent; 2. Subjects are in good health, without any clinical significant symptoms or laboratory test; 3. Having a body mass index between 19 and 28 kilogram per meter square (kg/m²); 4. Capable of giving written informed consent 5. Understanding and being willing to comply with the requirements of protocol, participate to complete the study; 6. Having recovered if received a surgery before . Exclusion criteria：

1. Allergic condition or having the history of allergic reactions to any drugs, pegylated products, or more than two substances;
2. Use of any medicine within 4 weeks or shorter than 5 half-lives;
3. Use of any medicine within 12 weeks, which is harm to any organ;
4. Participated in any other clinical trial within 12 weeks;
5. History of blood donation within 12 weeks;
6. History of glucose-6-phosphate dehydrogenase deficiency;
7. History of catalase deficiency;
8. Any significant disease, including but not limited to the following: digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, neuropsychiatry system, hematological system, immune system, metabolic system abnormity.
9. Abnormal significance clinical laboratory tests within 2 weeks such as routine blood test and urinalysis, blood chemistry, ECG.
10. Positive serology for hepatitis B surface antigen , or antibodies to hepatitis C, or HIV and syphilis;
11. Pregnancy, planning pregnancy, or breastfeeding;
12. Positive pregnancy test;
13. Male subject without effective contraception or his partner intend to be pregnant within 6 months;
14. History of mental disorder or disabilities legally;
15. History of alcohol abusing during the last 6 months;
16. More than 5 cigarettes per day during the last 6 months;
17. Positive drug abuse or alcohol test;
18. More than 1L of strong tea, coffee or caffeine drink per day;
19. Can't understand the content of informed consent form ;
20. Any condition, which investigators consider, is not fit for the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | baseline to 4 weeks
  incidence of adverse events
maximum tolerable dose | baseline to 4 weeks
  maximum tolerable dose

SECONDARY OUTCOMES:
peak plasma concentration | baseline to 4 weeks
  peak plasma concentration
area under the plasma concentration versus time curve | baseline to 4 weeks
  area under the plasma concentration versus time curve
level of serum uric acid | baseline to 4 weeks
  level of serum uric acid
Immunogenicity | baseline to 52 weeks
  anti-SSS11

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Shentu, Doctor, Principal Investigator — The First Affilicated Hospital Zhejiang University
Locations (1):
- The First Affilicated Hospital Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided